CLINICAL TRIAL: NCT01305356
Title: A Prospective, Randomized, Controlled, Multi-Center, Pivotal Human Clinical Trial to Evaluate the Safety and Effectiveness of Augment® Injectable Bone Graft Compared to Autologous Bone Graft as a Bone Regeneration Device in Hindfoot Fusions
Brief Title: Augment® Injectable Bone Graft Compared to Autologous Bone Graft as a Bone Regeneration Device in Hindfoot Fusions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioMimetic Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BMTI-2010-01; NCT01008891 (obsolete NCT alias)
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Degenerative Joint Disease; Congenital Deformity; Arthritis; Osteoarthritis; Rheumatoid Arthritis
Keywords: degenerative joint disease; DJD; joint fusion; hindfoot; congenital deformity; osteoarthritis; rheumatoid arthritis; post-traumatic arthritis; ankylosing spondylitis; Augment(tm) Injectable Bone Graft; autologous bone graft; autogenous bone graft; beta-TCP; bovine collagen; rhPDGF(bb)
MeSH Terms: conditions — Joint Diseases; Congenital Abnormalities; Arthritis; Osteoarthritis; Arthritis, Rheumatoid; Ankylosis; Spondylitis, Ankylosing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Augment® Injectable Bone Graft (Experimental): Standard rigid fixation + Augment® Injectable Bone Graft (beta-TCP/bovine collagen matrix + rhPDGF-BB)
  Interventions: Device: Augment® Injectable Bone Graft
- Autologous bone graft (Active Comparator): Standard Rigid Fixation + Autologous bone graft
  Interventions: Procedure: Autologous bone graft

INTERVENTIONS:
Device: Augment® Injectable Bone Graft — Implantation of up to 9cc of Augment® Injectable Bone Graft
  Arms: Augment® Injectable Bone Graft
Procedure: Autologous bone graft — Implantation of up to 9cc of autologous bone graft
  Arms: Autologous bone graft

SUMMARY:
STUDY OBJECTIVES:

To demonstrate equivalent clinical and radiologic outcomes as "gold standard" (Autologous Bone Graft) in a representative clinical model (hindfoot fusions)

STUDY HYPOTHESIS:

Augment® Injectable is an equivalent bone grafting substitute to autologous bone graft in applications as shown by superiority analysis for safety and non-inferiority analysis for effectiveness

STUDY RATIONALE:

To evaluate a fully synthetic bone graft material to facilitate fusion in conditions or injuries requiring bone graft in a representative clinical fusion model and thus the opportunity to provide equivalent union rates as Autologous Bone Graft without necessitating an additional invasive procedure to harvest the graft

DETAILED DESCRIPTION:
STUDY DESIGN:

Prospective, randomized, controlled, non-inferiority, multi-center trial

NUMBER OF STUDY CENTERS:

25

NUMBER OF SUBJECTS:

299 Subjects (see "Study Population"). The subject population included subjects enrolled in 3 separate Clinical Trials. (BMTI-2006-01, BMTI-2009-01, and BMTI-2010-01)

STUDY POPULATION:

Male and female subjects 18 years of age or older requiring a hindfoot fusion procedure involving a bone grafting procedure.

TREATMENT GROUPS:

Group I: Standard Rigid Fixation + Autologous Bone Graft Group II: Standard Rigid Fixation + Augment® Injectable Bone Graft

Subjects will be randomized in a 2:1 ratio (Augment® Injectable:Autologous Bone Graft).

ROUTE OF ADMINISTRATION:

Investigational device is manually implanted inside and around the fusion space to ensure Augment® Injectable Bone Graft (beta-TCP/bovine collagen matrix +rhPDGF-BB) or autologous bone graft is contained within the joint space

STUDY DURATION:

Twenty-four month follow-up post-surgery

ELIGIBILITY:
KEY INCLUSION CRITERIA:

* at least 18 years old and considered skeletally mature
* diagnosed with degenerative joint disease (DJD) affecting the hindfoot due to a congenital or acquired deformity, osteoarthritis, rheumatoid arthritis, post- traumatic arthritis or ankylosing spondylitis of the ankle, subtalar, calcaneocuboid, and/or talonavicular joints
* requires one of the following hindfoot fusion proceduress with supplemental bone graft/substitute: ankle fusion (tibiotalar), subtalar fusion (talocalcaneal), calcaneocuboid fusion, talonavicular fusion, triple arthrodesis (subtalar, talonavicular and calcaneocuboid joints) OR double fusions (any combination of any two of the following: subtalar, talonavicular and calcaneocuboid joints)
* fusion site able to be rigidly stabilized with no more than 3 screws across the fusion site

  * supplemental pins or staples allowed
  * supplemental screws external to the fusion site(s) allowed
* signed informed consent document, independent, ambulatory, and can comply with all post-operative evaluations and visits

KEY EXCLUSION CRITERIA:

* undergone previous fusion surgery at the proposed location, i.e., revision of a failed fusion
* more than one previous procedure at the involved joints
* retained hardware spanning the joint(s) intended for fusion
* procedure anticipated to require plate fixation (including claw plates), IM nails or more than 3 screws to achieve rigid fixation based on pre-op planning
* procedure expected to require more than 9cc of graft material based on pre-op planning
* procedure expected to require structural bone graft, allograft, bone graft substitute, platelet rich plasma (PRP) or bone marrow aspirate
* procedure expected to require a pantalar fusion, i.e., fusion of ankle plus all hindfoot joints (talonavicular, subtalar, and calcaneocuboid) or an ankle fusion in combination with any hindfoot fusion
* radiographic evidence of bone cysts, segmental defects or growth plate fracture near the fusion site that could negatively impact the proposed fusion procedure
* tested positive or been treated for a malignancy in the past or is suspected of having a malignancy or currently undergoing radio- or chemotherapy treatment for a malignancy anywhere in the body, whether adjacent to or distant from the proposed surgical site
* pre-existing sensory impairment, e.g., diabetics with baseline sensory impairment, which limits ability to perform objective functional measurements and may be at risk for complications

  - diabetics not sensitive to the 5.07 monofilament (Semmes-Weinstein) are to be excluded
* metabolic disorder known to adversely affect the skeleton other than primary osteoporosis or diabetes, e.g., renal osteodystrophy or hypercalcemia
* use of chronic medications known to affect the skeleton, e.g., glucocorticoid usage > 10mg/day
* pre-fracture neuromuscular or musculoskeletal deficiency which limits the ability to perform objective functional measurements
* physically or mentally compromised, e.g., current treatment for a psychiatric disorder, senile dementia, Alzheimer's disease, etc., to the extent that the Investigator judges the subject to be unable or unlikely to remain compliant
* allergic to yeast-derived products or bovine collagen or other bovine-sourced products
* received an investigational therapy within 30 days of proposed surgery or during the follow-up phase of the study
* is a prisoner, known or suspected transient or a history of drug/alcohol abuse within the 12 months prior to screening
* pregnant or intending to become pregnant within 12 months of the study procedure
* morbidly obese defined as BMI > 45 kg/m2
* currently has an acute infection at the surgical site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Roach, Study Director — Stryker Trauma and Extremities; Christopher DiGiovanni, MD, Principal Investigator — University Orthopaedics, Inc.
Locations (25):
- United States (20):
  - Tucson Orthopaedic Research Center, Tucson, Arizona
  - University of Arizona, Tucson, Arizona
  - California Pacific Medical Center, San Francisco, California
  - Illinois Bone & Joint Institute, Ltd., Glenview, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Union Memorial Hospital, Baltimore, Maryland
  - Mid Michigan Orthopaedic Institute, East Lansing, Michigan
  - Orthopaedic Associates of Michigan, PC, Grand Rapids, Michigan
  - Desert Orthopaedic Center, Las Vegas, Nevada
  - University of Medicine & Dentistry of New Jersey, Newark, New Jersey
  - Hospital for Special Surgery, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - OrthoCarolina, PA, Charlotte, North Carolina
  - Cleveland Clinic Orthopaedic, Cleveland, Ohio
  - Orthopedic Foot & Ankle Center, Columbus, Ohio
  - Health Research Institute, Inc., Oklahoma City, Oklahoma
  - The Rothman Institute, Philadelphia, Pennsylvania
  - Campbell Clinic / InMotion Orthopaedic Research Center, Memphis, Tennessee
  - Texas Health Research & Education Institute, Dallas, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
- Canada (5):
  - Life Mark Health Centre, Calgary, Alberta
  - St. Paul's Hospital, Vancouver, British Columbia
  - Queen Elizabeth II Health Services, Halifax, Nova Scotia
  - The Ottawa Hospital, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Result] Daniels TR, Younger AS, Penner MJ, Wing KJ, Le IL, Russell IS, Lalonde KA, Evangelista PT, Quiton JD, Glazebrook M, DiGiovanni CW. Prospective Randomized Controlled Trial of Hindfoot and Ankle Fusions Treated With rhPDGF-BB in Combination With a beta-TCP-Collagen Matrix. Foot Ankle Int. 2015 Jul;36(7):739-48. doi: 10.1177/1071100715576370. Epub 2015 Apr 6. PMID 25848134
- [Result] DiGiovanni CW, Lin SS, Baumhauer JF, Daniels T, Younger A, Glazebrook M, Anderson J, Anderson R, Evangelista P, Lynch SE; North American Orthopedic Foot and Ankle Study Group. Recombinant human platelet-derived growth factor-BB and beta-tricalcium phosphate (rhPDGF-BB/beta-TCP): an alternative to autogenous bone graft. J Bone Joint Surg Am. 2013 Jul 3;95(13):1184-92. doi: 10.2106/JBJS.K.01422. PMID 23824386

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A propensity score matching analysis was performed in order to identify a single set of investigational and control subjects derived from the datasets (BMTI-2006-01, BMTI-2009-01, BMTI-2010-01) that were comparable and could be evaluated for the purpose of assessing the safety and effectiveness of AUGMENT® Injectable.
Period: Overall Study
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Started | 132 | 167
Completed | 132 | 167
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft | Total
Number analyzed (Participants) | 132 | 167 | 299
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 97 | 109 | 206
  >=65 years | 35 | 58 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 81 | 143
  Male | 70 | 86 | 156
Affected Foot/Ankle [Count of Participants; unit: Participants]
  Ankle fusion | 31 | 46 | 77
  Subtalar fusion | 52 | 59 | 111
  Calcaneocuboid fusion | 3 | 0 | 3
  Talonavicular fusion | 6 | 9 | 15
  Double fusion | 21 | 17 | 38
  Triple arthordesis | 19 | 36 | 55
Ever smoked [Count of Participants; unit: Participants]
  No | 61 | 83 | 144
  Yes | 71 | 84 | 155

OUTCOME MEASURES:

1. Primary Outcome: Pain on Weight Bearing
Description: Subjects were asked to stand and report pain on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).
Time Frame: Baseline, 9, 12, 16, 24, 36, and 52 weeks
Population: Analysis conducted on patients at Baseline, 9, 12, 16, 24, 36, and 52 weeks time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Number analyzed (Participants) | 132 | 167
units on a scale
  Baseline: number analyzed (Participants) | 132 | 164
  Baseline | 71.0 (2.0) | 70.7 (1.8)
  Week 9: number analyzed (Participants) | 108 | 136
  Week 9 | 29.5 (2.9) | 28.2 (2.5)
  Week 12: number analyzed (Participants) | 124 | 154
  Week 12 | 26.8 (2.5) | 24.6 (2.2)
  Week 16: number analyzed (Participants) | 129 | 159
  Week 16 | 26.4 (2.4) | 24.4 (2.1)
  Week 24: number analyzed (Participants) | 128 | 160
  Week 24 | 25.1 (2.4) | 18.3 (2.1)
  Week 36: number analyzed (Participants) | 124 | 156
  Week 36 | 18.7 (2.3) | 15.8 (2.0)
  Week 52: number analyzed (Participants) | 124 | 157
  Week 52 | 16.6 (2.4) | 15.9 (2.1)

2. Secondary Outcome: Foot Function Index (FFI)
Description: The Foot Function Index (FFI) measures the impact of foot pathology on function in terms of pain, disability and activity restriction. The FFI is a self-administered index consisting of 23 items divided into 3 sub-scales all ranging from 0-100. To obtain a sub-scale score, the item scores for a sub-scale are totaled and then divided by the maximum total possible for all of the sub-scale items which the subject indicated were applicable. Any item marked as not applicable is excluded from the total possible. Sub-scales are an average of the completed ratings within that sub-scale. The total foot function score is an average of the three sub-scale scores and ranges from 0-100. Lower scores are indicative of better outcomes whereas higher scores indicate greater impairment.
Time Frame: Baseline, 9, 12, 16, 24, 36, and 52 weeks
Population: Analysis conducted on patients at Baseline, 9, 12, 16, 24, 36, and 52 weeks time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Number analyzed (Participants) | 132 | 167
units on a scale
  Baseline | 50.6 (1.6) | 50.0 (1.4)
  9 Weeks: number analyzed (Participants) | 126 | 157
  9 Weeks | 41.8 (1.7) | 45.0 (1.5)
  12 Weeks: number analyzed (Participants) | 126 | 161
  12 Weeks | 33.3 (1.8) | 34.5 (1.6)
  16 Weeks: number analyzed (Participants) | 127 | 162
  16 Weeks | 29.7 (2.0) | 28.0 (1.7)
  24 Weeks: number analyzed (Participants) | 129 | 164
  24 Weeks | 26.3 (1.8) | 19.8 (1.6)
  36 Weeks: number analyzed (Participants) | 124 | 159
  36 Weeks | 21.8 (1.8) | 16.7 (1.6)
  52 Weeks: number analyzed (Participants) | 123 | 160
  52 Weeks | 19.6 (1.9) | 16.9 (1.6)

3. Secondary Outcome: AOFAS Hindfoot and Ankle Score
Description: Subjects were asked to report pain, functionality and ability levels while the physician performed assessments based on alignment, abnormality, motion, and stability. The total score ranges from a low of zero to a high of 100, with subscales measuring pain (40 points), function (50 points), and alignment (10 points), with higher scores showing better outcomes.
Time Frame: Baseline, 9, 12, 16, 24, 36, and 52 weeks
Population: Analysis conducted on patients at Baseline, 9, 12, 16, 24, 36, and 52 weeks time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Number analyzed (Participants) | 132 | 167
units on a scale
  Baseline | 43.3 (1.5) | 43.6 (1.3)
  9 Weeks: number analyzed (Participants) | 126 | 155
  9 Weeks | 61.5 (1.1) | 61.5 (1.0)
  12 Weeks: number analyzed (Participants) | 124 | 162
  12 Weeks | 66.9 (1.3) | 66.6 (1.1)
  16 Weeks: number analyzed (Participants) | 129 | 163
  16 Weeks | 69.9 (1.3) | 71.2 (1.1)
  24 Weeks: number analyzed (Participants) | 129 | 164
  24 Weeks | 73.4 (1.5) | 75.5 (1.3)
  36 Weeks: number analyzed (Participants) | 124 | 160
  36 Weeks | 77.5 (1.5) | 78.9 (1.3)
  52 Weeks: number analyzed (Participants) | 125 | 160
  52 Weeks | 79.5 (1.6) | 79.3 (1.4)

4. Secondary Outcome: Fusion Site Pain
Description: Subjects were asked to report current pain level at the fusion site on a 100 mm Visual Analog Scale (with 0 being no pain and 100 being worst pain imaginable).
Time Frame: Baseline, 9, 12, 16, 24, 36, and 52 weeks
Population: Analysis conducted on patients at Baseline, 9, 12, 16, 24, 36, and 52 weeks time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Number analyzed (Participants) | 132 | 167
units on a scale
  Baseline | 51.4 (2.4) | 50.4 (2.1)
  Week 9: number analyzed (Participants) | 126 | 158
  Week 9 | 20.5 (2.1) | 15.4 (1.8)
  Week 12: number analyzed (Participants) | 126 | 162
  Week 12 | 18.9 (2.1) | 17.8 (1.8)
  Week 16: number analyzed (Participants) | 129 | 162
  Week 16 | 21.7 (2.2) | 18.9 (2.0)
  Week 24: number analyzed (Participants) | 129 | 164
  Week 24 | 20.9 (2.2) | 15.3 (1.9)
  Week 36: number analyzed (Participants) | 124 | 159
  Week 36 | 17.4 (2.1) | 12.4 (1.8)
  Week 52: number analyzed (Participants) | 125 | 160
  Week 52 | 15.8 (2.2) | 12.6 (1.9)

5. Secondary Outcome: SF-12 Physical Component Score
Description: The SF-12 Physical Component Score is a validated quality of life metric with a minimum of zero and a maximum of 100, with higher scores denoting higher quality of life.
Time Frame: Baseline, 9, 12, 16, 24, 36, and 52 weeks
Population: Analysis conducted on patients at Baseline, 12, 16, 24, 36, and 52 weeks time points.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
Number analyzed (Participants) | 132 | 167
units on a scale
  Baseline | 30.8 (0.8) | 30.8 (0.7)
  Week 12: number analyzed (Participants) | 126 | 158
  Week 12 | 36.9 (0.8) | 36.3 (0.7)
  Week 16: number analyzed (Participants) | 128 | 162
  Week 16 | 37.9 (0.8) | 39.0 (0.7)
  Week 24: number analyzed (Participants) | 129 | 164
  Week 24 | 40.3 (0.9) | 42.2 (0.7)
  Week 36: number analyzed (Participants) | 124 | 159
  Week 36 | 42.1 (0.9) | 44.5 (0.8)
  Week 52: number analyzed (Participants) | 123 | 160
  Week 52 | 42.9 (0.9) | 45.5 (0.8)

ADVERSE EVENTS:
Time Frame: Patients were assessed through study completion scheduled at 52 weeks following surgery.
Arm/Group | Augment® Injectable Bone Graft | Autologous Bone Graft
All-Cause Mortality (participants affected / at risk) | 0/132 | 0/167
Serious Adverse Events (participants affected / at risk) | 20/132 | 35/167
Other Adverse Events (participants affected / at risk) | 116/132 | 135/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Augment® Injectable Bone Graft (N=132) | Autologous Bone Graft (N=167)
Anemia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 | 1
gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Megacolon (Gastrointestinal disorders) | 0 | 1
Impaired healing (General disorders) | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Ureteric injury (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 3
Hematoma (Vascular disorders) | 1 | 0
Pulmonary embolism (Vascular disorders) | 0 | 1
Device related infection (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 1
Wound infection (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Augment® Injectable Bone Graft (N=132) | Autologous Bone Graft (N=167)
Nausea (Gastrointestinal disorders) | 20 | 12
Feeling Hot (General disorders) | 16 | 6
Local Swelling (General disorders) | 27 | 13
Medical Device Discomfort (General disorders) | 7 | 3
Pyrexia (General disorders) | 7 | 2
Tenderness (General disorders) | 22 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 28 | 19
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 7
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 7 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 35
Headache (Nervous system disorders) | 7 | 2
Hypoaesthesia (Nervous system disorders) | 10 | 10
Anemia (Blood and lymphatic system disorders) | 1 | 2
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 4 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Chest discomfort (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Syncope (Cardiac disorders) | 1 | 0
Congenital foot malformation (Congenital, familial and genetic disorders) | 0 | 1
Talipes (Congenital, familial and genetic disorders) | 0 | 1
Labyrinthitis (Ear and labyrinth disorders) | 1 | 0
Otitis media (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 1
Diabetes mellitus (Endocrine disorders) | 1 | 0
Diabetic neuropathy (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 2 | 0
Cataract (Eye disorders) | 0 | 1
Chalazion (Eye disorders) | 1 | 0
Eye pain (Eye disorders) | 1 | 0
Optic disc disorder (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 4
Diarrhea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Megacolon (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Procedural nausea (Gastrointestinal disorders) | 0 | 1
Tooth infection (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 4 | 8
Administration site pain (General disorders) | 1 | 0
Chills (General disorders) | 4 | 1
Drug withdrawal syndrome (General disorders) | 0 | 1
Impaired healing (General disorders) | 6 | 5
Inflammation (General disorders) | 1 | 1
Necrosis (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 1 | 6
Pain (General disorders) | 2 | 1
Soft tissue inflammation (General disorders) | 0 | 1
Swelling (General disorders) | 1 | 1
Ulcer (General disorders) | 0 | 1
Gallbladder pain (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 5
Cellulitis (Infections and infestations) | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 4 | 3
Influenza (Infections and infestations) | 1 | 2
Kidney infection (Infections and infestations) | 0 | 2
Localised infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 6
Onychomycosis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 2
Staphylococcal infection (Infections and infestations) | 3 | 2
Tooth abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 3 | 2
Viral labyrinthitis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 2
Arteriovenous graft site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Blister (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 0 | 1
Burns third degree (Injury, poisoning and procedural complications) | 0 | 1
Bursa injury (Injury, poisoning and procedural complications) | 0 | 1
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 4 | 3
Corneal abrasion (Injury, poisoning and procedural complications) | 1 | 0
Device related infection (Injury, poisoning and procedural complications) | 0 | 1
Eschar (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 5 | 5
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 2
Graft complication (Injury, poisoning and procedural complications) | 0 | 8
Graft infection (Injury, poisoning and procedural complications) | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 0 | 3
Limb injury (Injury, poisoning and procedural complications) | 0 | 2
Medical device complication (Injury, poisoning and procedural complications) | 3 | 3
Medical device pain (Injury, poisoning and procedural complications) | 0 | 6
Medical device site reaction (Injury, poisoning and procedural complications) | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 1 | 0
Necrotic preservation injury of graft (Injury, poisoning and procedural complications) | 1 | 0
Nerve compression (Injury, poisoning and procedural complications) | 0 | 1
Open wound (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 2
Peroneal nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Post procedural cellulitis (Injury, poisoning and procedural complications) | 0 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural oedema (Injury, poisoning and procedural complications) | 0 | 1
Postoperative wound infection (Injury, poisoning and procedural complications) | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 2
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1
Stress fracture (Injury, poisoning and procedural complications) | 2 | 2
Superficial injury of eye (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 1
Wound decomposition (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 5 | 2
Wound infection (Injury, poisoning and procedural complications) | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 2
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1
Respiratory rate decreased (Investigations) | 0 | 1
Urine analysis (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 0 | 1
Oedema (Metabolism and nutrition disorders) | 1 | 0
Oedema peripheral (Metabolism and nutrition disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Arthritis infective (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bunion (Musculoskeletal and connective tissue disorders) | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 | 2
Gout (Musculoskeletal and connective tissue disorders) | 0 | 3
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint crepitation (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint dislocation (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint sprain (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 2
Monarthritis (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 | 3
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 3
Synovial cyst (Musculoskeletal and connective tissue disorders) | 2 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 2
Bone cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Complex regional pain syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 0
Hyperpathia (Nervous system disorders) | 1 | 0
Insomnia (Nervous system disorders) | 3 | 3
Neuralgia (Nervous system disorders) | 2 | 3
Neuritis (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 6
Paraesthesia (Nervous system disorders) | 2 | 1
Peroneal nerve injury (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 1 | 1
Sinus headache (Nervous system disorders) | 1 | 0
Tarsal tunnel syndrome (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 1
Urinary incontinence (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Vomiting in pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Mood altered (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Incontinence (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 2
Ureteric injury (Renal and urinary disorders) | 0 | 1
Ureteric stenosis (Renal and urinary disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 2 | 4
Urinary tract infection (Renal and urinary disorders) | 2 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 2 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Application site vesicles (Skin and subcutaneous tissue disorders) | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 6 | 3
Blood blister (Skin and subcutaneous tissue disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Eschar (Skin and subcutaneous tissue disorders) | 1 | 1
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0
Excoriation (Skin and subcutaneous tissue disorders) | 0 | 1
Hypoaesthesia facial (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomycosis (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 4
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1
Scar pain (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Splinter haemorrhages (Skin and subcutaneous tissue disorders) | 1 | 0
Bladder neoplasm surgery (Surgical and medical procedures) | 0 | 1
Cast application (Surgical and medical procedures) | 0 | 1
Endodontic procedure (Surgical and medical procedures) | 2 | 0
Gastric banding (Surgical and medical procedures) | 0 | 1
Incisional drainage (Surgical and medical procedures) | 0 | 1
Mole excision (Surgical and medical procedures) | 0 | 1
Splint application (Surgical and medical procedures) | 1 | 0
Ureteral stent removal (Surgical and medical procedures) | 0 | 1
Wound drainage (Surgical and medical procedures) | 3 | 2
Aneurysm (Vascular disorders) | 1 | 0
Aortic arteriosclerosis (Vascular disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 0 | 2
Deep vein thrombosis (Vascular disorders) | 3 | 4
Haematoma (Vascular disorders) | 2 | 1
Haemorrhage (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 2
Procedural hypertension (Vascular disorders) | 0 | 1
Pulmonary embolism (Vascular disorders) | 0 | 1
Rectal haemorrhage (Vascular disorders) | 1 | 0
Varicose vein (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes